CLINICAL TRIAL: NCT00904696
Title: Assessment of Tolerability & Effectiveness of Progut in Treatment of Irritable Bowel Syndrome
Brief Title: Tolerability and Effectiveness of Progut in Treatment of Irritable Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Medicine, Professor & Senior Consultant Gastroenterologist, Ho Khek Yu, National University Hospital, Singapore
Other Study IDs: E/08/532
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable bowel syndrome; probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Irritable bowel syndrome (IBS) is a very common chronic functional gastrointestinal disorder characterised by abdominal pain/discomfort, bloating and alterations in bowel function. This condition significantly impairs quality of life and places a large burden on health care resources. Existing therapies for IBS are far from being satisfactory and new therapies are being constantly sought.

The pathogenesis of IBS remains unclear. Imbalance in the intestinal microbiota is considered to be one important etiologic factor for IBS. That some probiotics are effective in the prevention and treatment of IBS supports this idea.

Progut is a synbiotic: a combination of probiotics and prebiotics. Probiotics are viable beneficial bacteria that are normally present in a healthy digestive tract. Each capsule of Progut contains 9 billion viable bacteria from 8 different strains that are characteristics of a healthy normal gut microflora: Lactobacillus (L. acidophilus, L. casei, L. lactis, and L. bulgaricus); Bifidobacterium (B. longum, B. infantis and B. bifidum); and Streptococcus thermophilus at time of manufacturing. To ensure survival of these bacteria, Progut is encapsulated and enteric-coated.

The primary objective is to evaluate the tolerability of Progut treatment 1-3 capsules/day in patients with irritable bowel syndrome under the same conditions as those likely to be encountered in a standard general clinical practice or outpatient clinic.

The rationale for this study is to obtain tolerability data in patients with IBS in the Singapore. The secondary objectives are to evaluate the patients' satisfaction and symptom improvement with Progut treatment.

DETAILED DESCRIPTION:
This will be an open-label, single arm post marketing surveillance study involving an active treatment period of a minimum 3-week and a maximum 12-week duration. Treatment with Progut will be at the discretion of the attending doctor and decision is independent of this study. This study will only recruit patients following the prescription of Progut and follow them up for upto a maximum of 12 weeks.

At Visit 1 (Day 1), the eligible patients will receive a prescription for Progut from their physician. Depending on the discretion of the attending physician, they will be prescribed Progut for treatment duration lasting 3 to 12 weeks. Safety of Progut under normal clinical use will be assessed at the end of this period. Perception of effectiveness, and tolerability of treatment will be assessed on Day 8-15 using a phone interview. On Visit 2 (any time between Day 22 to 85, depending on duration of treatment given and schedule of their follow-up visit arranged by the attending physician), the patient will be evaluated for symptomatic improvement, perception of effectiveness, tolerability and satisfaction with treatment, following which he/she will formally exit the study.

This study design was chosen with the aim of recruiting rapidly a large cohort of patients representative of the population being prescribed Progut. A total of 50 patients will be included to allow for an assessment of patient's tolerability of Progut, as well as satisfaction and perception of effectiveness and symptom response in the Singapore population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above with IBS diagnosed by the presence of the following symptoms:

  * abdominal pain,
  * bloating and constipation in whom organic pathology has been excluded
* All patients would have had endoscopy done in the past 3 years to exclude organic lower gastrointestinal pathology.
* All patients would have been prescribed Progut (1-3 capsules per day)by their physicians.

Exclusion Criteria:

* Women who are pregnant, intending to become pregnant or breastfeeding.
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Immunocompromised patients
* Hypersensitivity to Progut

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study subjects will be patients aged 18 years and older, diagnosed with IBS by their own physicians, and determined to be eligible to receive a prescription for Progut. In addition, they must satisfy the inclusion criteria stated below, be able to communicate well, provide written informed consent required by local regulations and willing to participate in the entire study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is patient's tolerance with the treatment. | 3-12 weeks

SECONDARY OUTCOMES:
Secondary endpoints are the resolution of gastrointestinal symptoms as assessed by a symptom questionnaire, patient's perception of effectiveness of the treatment and their overall satisfaction with the treatment. | 3-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Khek Yu Ho, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] O'Mahony L, McCarthy J, Kelly P, Hurley G, Luo F, Chen K, O'Sullivan GC, Kiely B, Collins JK, Shanahan F, Quigley EM. Lactobacillus and bifidobacterium in irritable bowel syndrome: symptom responses and relationship to cytokine profiles. Gastroenterology. 2005 Mar;128(3):541-51. doi: 10.1053/j.gastro.2004.11.050. PMID 15765388
- [Background] Malinen E, Rinttila T, Kajander K, Matto J, Kassinen A, Krogius L, Saarela M, Korpela R, Palva A. Analysis of the fecal microbiota of irritable bowel syndrome patients and healthy controls with real-time PCR. Am J Gastroenterol. 2005 Feb;100(2):373-82. doi: 10.1111/j.1572-0241.2005.40312.x. PMID 15667495